CLINICAL TRIAL: NCT03669744
Title: Regional Anesthesia in Refractory Trigeminal Neuralgia: 21 Cases Reported to the Limoges University Hospital
Acronym: TRINEB ONE
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_0004 (TRINEB ONE)
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-07

CONDITIONS: Trigeminal Neuralgia
Keywords: chronic pain; trigeminal neuralgia; regional anesthesia; trigeminal nerve block
MeSH Terms: conditions — Trigeminal Neuralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with trigeminal neuralgia resistant: a telephone survey will be conducted at 21 patients with trigeminal neuralgia resistant to usual treatments, according to the ICHD-3β criteria treating by one or more trigeminal nerve blocks at the peri operative pain management center of Limoges University Hospital between 2014 and 2018
  Interventions: Other: telephone survey

INTERVENTIONS:
Other: telephone survey — a telephone survey will be conducted at 21 patients with trigeminal neuralgia resistant to usual treatments, according to the ICHD-3β criteria treating by one or more trigeminal nerve blocks at the peri operative pain management center of Limoges University Hospital between 2014 and 2018.

SUMMARY:
Trigeminal neuralgia is defined according to the third edition of the International Classification of Headache Disorders (ICHD-3) criteria. Chronic pain can have a major impact on the quality of life. First-line treatments are anti-epileptics, and surgical treatments are also possible according to several approaches. Sometimes the pain is resistant to these therapies. In this indication, sensory blocks may have a therapeutic impact but their place is not clear. In France, there are formalized expert recommendations on "loco regional analgesia and chronic pain", from 2013. Several adjuvants to local anesthetics have been studied for acute and chronic pain. CLONIDINE and DEXAMETHASONE are of greatest interest in increasing block duration and reducing opioid consumption. The investigators report the case of 21 patients, treated by a trigeminal block from 2014 to 2018, suffering from a resistant trigeminal neuralgia. After a first consultation, the diagnosis is confirmed, an information is done and an appropriate support is established. The sensory block is performed as an outpatient care. It consists in a peri-neural injection of a mixture of LEVOBUPIVACAINE 5%, CORTIVAZOL 3.75mg / 1.5mL (or BETAMETHASONE 7mg / 1ml) and CLONIDINE (1μg / kg). Standard precautions are respected and patients are monitored in the recovery room after the procedure. The efficacity is evaluated before the exit and a follow-up is done within 15 days. The level of satisfaction expressed by the patients seems to be globally high. The investigators wish to evaluate statistically the impact of the trigeminal blocks, in terms of improvement of the quality of life. This retrospective study, by its procedure, does not change the management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with trigeminal neuralgia resistant to usual treatments, according to the ICHD-3β criteria
* treating by one or more trigeminal nerve blocks
* at the peri operative pain management center of Limoges University Hospital
* between 2014 and 2018

Exclusion Criteria:

* Not consent
* Another type of facial block during the previous year.
* Unavailable medical data
* Deceased patient

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with trigeminal neuralgia resistant to usual treatments, according to the ICHD-3β criteria treating by one or more trigeminal nerve blocks at the peri operative pain management center of Limoges University Hospital between 2014 and 2018.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Change of the quality of life from baseline to day 15 after baseline | Day 0, Day 15
  Percentage of patients with improvement of more than 50% in quality of life, mesured with the 'Medical Outcome Study Short Form 12', from baseline (day 0 = just before the block) to day 15. The questionnaire consists of 12 items questioned weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better health.

SECONDARY OUTCOMES:
Change in pain level just before and after the block assessed by a numerical scoring scale | Day 0, Day 15
  Average value of the Numerical Rating Scale immediately before, after and at day 15 after the block. Zero represents 'no pain at all' whereas ten represents 'the worst pain ever possible'
Neuropathic criteria of pain just before and after the block assessed by DN4 | Day 0
  Average value of the DN4 score before and after the block. DN4 questionnaire helps estimate the likelihood of neuropathic pain. The maximum score is 10. The threshold value for the diagnosis of neuropathic pain is 4.
Duration of the block | Day 0
  Number of days before covering an VAS justifying a new block
Patient overall satisfaction assessed by a Numerical Rating Scale. | Day 0
  Average value of the Numerical Rating Scale. Zero represents 'not at all satisfied' whereas ten represents 'very satisfied'.
Impact on analgesics consumption assessed by the dosage of analgesics | Day 0
  doses of analgesics compared to those usually delivered
Side effects | Day 0
  To list side effects
Return to work | Day 0
  For the patients concerned: yes / no
Return to hobbies | Day 0
  For the patients concerned: yes / no

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie NATHAN-DENIZOT, PU-PH, Principal Investigator — University Hospital, Limoges
Locations (1):
- University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No